CLINICAL TRIAL: NCT06180512
Title: Randomized Clinical Trial to Analyze the Efficacy of Acute Intake of Different Doses of a β-alanine Supplement on Performance in Recreational Cross-country Road Cyclists
Brief Title: Study to Analyze the Efficacy of Acute Intake With a β-alanine Supplement in Recreational Cyclists
Acronym: B-AC1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Francisco Javier López Román, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: UCAMCFE-00029
Record Dates: First submitted 2023-12-02; First posted 2023-12-22 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2023-11

CONDITIONS: Beta Alanine Supplementation
Keywords: Acute effect; Beta Alanine
MeSH Terms: interventions — beta-Alanine; Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Beta Alanine high dose (Experimental): Consumption for 1 day.
  Interventions: Dietary Supplement: Beta Alanine high dose
- Beta Alanine low dose (Experimental): Consumption for 1 day.
  Interventions: Dietary Supplement: Beta Alanine low dose
- Control group (Placebo Comparator): Consumption for 1 day.
  Interventions: Dietary Supplement: Control group

INTERVENTIONS:
Dietary Supplement: Beta Alanine high dose — 4 intakes of 5 g of beta alanine every 1 hour and 15 minutes.
  Arms: Beta Alanine high dose
Dietary Supplement: Beta Alanine low dose — 4 intakes of 2.5 g of beta alanine every 1 hour and 15 minutes.
  Arms: Beta Alanine low dose
Dietary Supplement: Control group — 4 intakes of 2.5 g of wheat semolina every 1 hour and 15 minutes.
  Arms: Control group

SUMMARY:
Randomized, controlled, double-blind, single-center, double-blind clinical trial with three parallel arms depending on the product consumed (experimental product dose 1 and dose 2 and placebo product) to measure the efficacy of a sustained release beta alanine on physiological physical performance efficacy in recreational cyclists.

DETAILED DESCRIPTION:
Subjects meeting the selection criteria will be randomly assigned to each of the study groups (investigational product dose 1 or dose 2, or placebo, depending on the group to which they have been assigned).

The product to be consumed is beta alanine. Participants will consume the product for 1 day. They will have to take four intakes every hour and a quarter, on the same day.

The study subjects will have to make 2 visits to the laboratory. In the first one, they will have to perform a 10-minute time trial, without consumption. In the second visit, they will perform the same performance test but with acute consumption of the product. Their physical and physiological performance will be evaluated.

The two tests will be separated by 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Male cyclists with more than two years of cycling experience.
* Perform tests without fatigue.
* Road bike training at least twice a week.

Exclusion Criteria:

* Participants with chronic illness.
* Have a long-term injury that prevents you from training in the previous month.
* Inability to understand informed consent.
* Have consumed beta alanine in the three years prior to the start of the study.
* Consumption of other supplements that may alter performance.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2023-12-04 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2024-01-22 (Actual)

PRIMARY OUTCOMES:
Power | It will be measured on two different occasions. Day one and seven days later with acute consumption of product.
  Physical performance is measured by direct variables evaluated by the power roller (average power, maximum power, etc.).
Distance covered | It will be measured on two different occasions. Day one and seven days later with acute consumption of product.
  Physical performance is measured by direct variables evaluated by the power roller.

SECONDARY OUTCOMES:
Fatigue | Change of baseline rate of perceived exertion at seven days
  Rate of perceived exertion, assessed by the 10-point modified Borg Scale.
Paresthesia test | It will be measured on two different occasions. on day 1 (before consumption) and seven days after (after consumption).
  Visual analogue scale (1-10)
Microcapillary blood | It will be measured on two different occasions. Day one and seven days later.
  This test provides biochemical variables (ABL90FLEX) with 70 ml of capillary blood (Na, K, Glucose, Lactate, etc). It is used to evaluate the effort made by the cyclist.
Lactate | It will be measured on two different occasions. Day one and seven days later.
  Lactate levels will be measured using the Lactate Pro
Heart Rate | It will be measured on two different occasions. Day one and seven days later.
  The heart rate will be evaluated by means of a heart rate strap.

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Murcia, Murcia, Spain